CLINICAL TRIAL: NCT04586920
Title: A Phase 1, Randomized, Participant-and Investigator-Blind, Placebo-Controlled, Single-and Multiple-Ascending Dose, Drug-Drug Interaction and Food Effect Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3509754 in Healthy Non-Japanese and Japanese Participants
Brief Title: A Study of LY3509754 in Healthy Non-Japanese and Japanese Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to safety findings
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17797; J3D-MC-FNAA (Other: Eli Lilly and Company); 2020-003957-30 (EudraCT Number)
Record Dates: First submitted 2020-10-13; First posted 2020-10-14 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- LY3509754 - Part A (Experimental): Escalating doses of 10, 30, 100, 300, 1000, and 2000 milligrams (mg) of LY3509754 were administered orally.
  Interventions: Drug: LY3509754
- Placebo - Part A (Placebo Comparator): Placebo was administered orally.
  Interventions: Drug: Placebo
- LY3509754 plus Itraconazole - Part B (Experimental): 10 mg of LY3509754 and 200 mg of Itraconazole were administered orally.
  Interventions: Drug: LY3509754; Drug: Itraconazole
- Placebo plus Itraconazole - Part B (Placebo Comparator): Placebo and 200 mg Itraconazole were administered orally.
  Interventions: Drug: Placebo; Drug: Itraconazole
- LY3509754 plus Midazolam - Part C (Experimental): Multiple doses of LY3509754 (100, 300, and 1000 mg) were administered orally. Some participants also received 1.2 mg midazolam orally.
  Interventions: Drug: LY3509754; Drug: Midazolam
- Placebo plus Midazolam - Part C (Placebo Comparator): Multiple doses of placebo were administered orally. Some participants also received 1.2 mg midazolam orally.
  Interventions: Drug: Placebo; Drug: Midazolam
- LY3509754 (Japanese) - Part D (Experimental): Multiple doses of LY3509754 (400 and 1000 mg) were administered orally to Japanese participants.
  Interventions: Drug: LY3509754
- Placebo (Japanese) - Part D (Placebo Comparator): Placebo was administered orally to Japanese participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3509754 — Administered orally
  Arms: LY3509754 (Japanese) - Part D; LY3509754 - Part A; LY3509754 plus Itraconazole - Part B; LY3509754 plus Midazolam - Part C
Drug: Placebo — Administered orally
  Arms: Placebo (Japanese) - Part D; Placebo - Part A; Placebo plus Itraconazole - Part B; Placebo plus Midazolam - Part C
Drug: Itraconazole — Administered orally
  Arms: LY3509754 plus Itraconazole - Part B; Placebo plus Itraconazole - Part B
Drug: Midazolam — Administered orally
  Arms: LY3509754 plus Midazolam - Part C; Placebo plus Midazolam - Part C

SUMMARY:
The main purpose of this study in healthy participants is to learn more about the safety of LY3509754 and any side effects that might be associated with it. Blood tests will be performed to check how much LY3509754 gets into the bloodstream and how long it takes the body to eliminate it.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history and physical examination.
* Body mass index (BMI) within the range of 18 to 35 kilograms per meter squared (kg/m²) in Parts A, B, and C. In Part D (Japanese participants), body weight between 50 and 85 kg and BMI within the range of 18 to 28 kg/m².

Exclusion Criteria:

* Have previously completed or withdrawn from this study or any other study investigating LY3509754, and have previously received LY3509754.
* Women of childbearing potential are excluded from the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Covance Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Datta-Mannan A, Regev A, Coutant DE, Dropsey AJ, Foster J, Jones S, Poorbaugh J, Schmitz C, Wang E, Woodman ME. Safety, Tolerability, and Pharmacokinetics of an Oral Small Molecule Inhibitor of IL-17A (LY3509754): A Phase I Randomized Placebo-Controlled Study. Clin Pharmacol Ther. 2024 May;115(5):1152-1161. doi: 10.1002/cpt.3185. Epub 2024 Jan 31. PMID 38294091

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - Placebo (Fasted): Participants received single oral dose of placebo under fasting condition.
- Part A - Placebo (Fed): Participants received single oral dose of placebo under fed condition.
- Part A - 10 Milligram (mg) LY3509754 (Fasted): Participants received a single oral dose of 10 mg LY3509754 under fasting condition.
- Part A - 30 mg LY3509754 (Fasted): Participants received a single oral dose of 30 mg LY3509754 under fasting condition.
- Part A - 100 mg LY3509754 (Fasted): Participants received a single oral dose of 100 mg LY3509754 under fasting condition.
- Part A - 300 mg LY3509754 (Fasted and Fed): Participants received a single oral dose of 300 mg LY3509754 under fasting condition. There was a washout period of at least 5 days. Participants received a single oral dose of 300 mg LY3509754 under fed condition.
- Part A - 1000 mg LY3509754 (Fasted): Participants received a single oral dose of 1000 mg LY3509754 under fasting condition.
- Part A - 2000 mg LY3509754 (Fasted): Participants received a single oral dose of 2000 mg LY3509754 under fasting condition.
- Part B - Placebo + 200 mg Itraconazole (Day 10): Participants received a single oral dose of placebo on Day 1 followed by daily doses of 200 mg itraconazole as oral solution for 10 days twice daily (BID) on Day 4 and once daily (QD) from Days 5 through 13. Participants received a single oral dose of placebo on Day 10.
- Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10): Participants received a single oral dose of 10 mg LY3509754 on Day 1 followed by daily doses of 200 mg itraconazole as oral solution for 10 days BID on Day 4 and QD from Days 5 through 13. Participants received a single oral dose of placebo on Day 10.
- Part C - QD [Cohorts 1 and 3]; Part D (Japanese) - Placebo QD: Participants received oral doses of placebo QD for 14 Days.
- Part C - 100 mg LY3509754 QD [Cohort 1]: Participants received oral doses of 100 mg LY3509754 QD for 14 Days.
- Part C - Placebo QD + 1.2 mg Midazolam [Cohort 2]: Participants received a single dose of 1.2 mg midazolam given as oral solution on Day -2 followed by oral doses of placebo QD from Day 1 to 15. Participants then received a single dose of 1.2 mg midazolam given as oral solution on Day 15.
- Part C - 300 mg LY3509754 QD + 1.2 mg Midazolam [Cohort 2]: Participants received a single dose of 1.2 mg midazolam given as oral solution on Day -2 followed by oral doses of 300 mg LY3509754 QD from Day 1 to 15. Participants then received a single dose of 1.2 mg midazolam given as oral solution on Day 15.
- Part C - 1000 mg LY3509754 QD [Cohort 3]; Part D (Japanese) - 1000 mg LY3509754 QD: Participants received oral doses of 1000 mg LY3509754 QD for 14 Days.
- Part D (Japanese) - 400 mg LY3509754 QD: Participants received oral doses of 400 mg LY3509754 QD for 14 Days.
Period: Overall Study
Arm/Group | Part A - Placebo (Fasted) | Part A - Placebo (Fed) | Part A - 10 Milligram (mg) LY3509754 (Fasted) | Part A - 30 mg LY3509754 (Fasted) | Part A - 100 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fasted and Fed) | Part A - 1000 mg LY3509754 (Fasted) | Part A - 2000 mg LY3509754 (Fasted) | Part B - Placebo + 200 mg Itraconazole (Day 10) | Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10) | Part C - QD [Cohorts 1 and 3] | Part C - 100 mg LY3509754 QD [Cohort 1] | Part C - Placebo QD + 1.2 mg Midazolam [Cohort 2] | Part C - 300 mg LY3509754 QD + 1.2 mg Midazolam [Cohort 2] | Part C - 1000 mg LY3509754 QD [Cohort 3] | Part D (Japanese) - Placebo QD | Part D (Japanese) - 400 mg LY3509754 QD | Part D (Japanese) - 1000 mg LY3509754 QD
Started | 10 | 2 | 6 | 6 | 6 | 9 | 6 | 6 | 3 | 8 | 4 | 6 | 2 | 8 | 6 | 4 | 6 | 6
Received At Least One Dose of Study Drug | 10 | 2 | 6 | 6 | 6 | 9 | 6 | 6 | 3 | 8 | 4 | 6 | 2 | 8 | 6 | 4 | 6 | 6
Completed | 10 | 2 | 6 | 6 | 6 | 9 | 5 | 4 | 3 | 6 | 4 | 5 | 2 | 7 | 6 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part A - 10 mg LY3509754 (Fasted): Participants received a single oral dose of 10 mg LY3509754 under fasting condition.
- Part B - Placebo + 200 mg Itraconazole (Day 10): Participants received a single oral dose of placebo on Day 1 followed by daily doses of 200 mg itraconazole as oral solution for 10 days BID on Day 4 and QD from Days 5 through 13. Participants received a single oral dose of placebo on Day 10.
- Part C - Placebo QD [Cohorts 1 and 3]; Part D (Japanese) - Placebo QD: Participants received oral doses of placebo QD for 14 Days.
- Total: Total of all reporting groups
Arm/Group | Part A - Placebo (Fasted) | Part A - Placebo (Fed) | Part A - 10 mg LY3509754 (Fasted) | Part A - 30 mg LY3509754 (Fasted) | Part A - 100 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fasted and Fed) | Part A - 1000 mg LY3509754 (Fasted) | Part A - 2000 mg LY3509754 (Fasted) | Part B - Placebo + 200 mg Itraconazole (Day 10) | Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10) | Part C - Placebo QD [Cohorts 1 and 3] | Part C - 100 mg LY3509754 QD [Cohort 1] | Part C - Placebo QD + 1.2 mg Midazolam [Cohort 2] | Part C - 300 mg LY3509754 QD + 1.2 mg Midazolam [Cohort 2] | Part C - 1000 mg LY3509754 QD [Cohort 3] | Part D (Japanese) - Placebo QD | Part D (Japanese) - 400 mg LY3509754 QD | Part D (Japanese) - 1000 mg LY3509754 QD | Total
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 6 | 9 | 6 | 6 | 3 | 8 | 4 | 6 | 2 | 8 | 6 | 4 | 6 | 6 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (13.0) | 43.5 (3.5) | 43.8 (16.1) | 43.8 (11.0) | 52.0 (10.4) | 52.9 (13.3) | 56.8 (4.6) | 42.0 (14.3) | 33.3 (6.8) | 42.6 (9.4) | 44.0 (8.5) | 43.2 (15.3) | 38.0 (2.8) | 46.5 (16.1) | 48.2 (12.2) | 52.5 (11.9) | 54.0 (7.5) | 50.0 (9.1) | 47.45 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 1 | 1 | 3 | 3 | 2 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 1 | 2 | 2 | 27
  Male | 7 | 2 | 4 | 5 | 5 | 6 | 3 | 4 | 3 | 8 | 3 | 4 | 1 | 5 | 6 | 3 | 4 | 4 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 1 | 4 | 4 | 5 | 0 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 26
  Not Hispanic or Latino | 9 | 2 | 4 | 5 | 5 | 5 | 2 | 1 | 3 | 6 | 3 | 3 | 1 | 8 | 5 | 4 | 6 | 6 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 2 | 2 | 3 | 3 | 3 | 2 | 1 | 5 | 3 | 3 | 2 | 2 | 1 | 4 | 2 | 0 | 0 | 0 | 38
  White | 7 | 0 | 3 | 2 | 3 | 6 | 4 | 1 | 0 | 4 | 2 | 4 | 1 | 4 | 3 | 0 | 0 | 0 | 44
  More than one race | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 2 | 6 | 6 | 6 | 9 | 6 | 6 | 3 | 8 | 4 | 6 | 2 | 8 | 6 | 4 | 6 | 6 | 104

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any adverse event (AE) from the study that results in 1 of the following: Death, initial or prolonged inpatient hospitalization, a life-threatening experience (i.e., immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect, important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent 1 of the other outcomes listed in the definition above.
  The number of participants with one or more SAEs considered by the investigator to be related to study drug administration is reported here. A summary of SAEs and other non-serious AEs, regardless of causality, will be reported in the Reported Adverse Events module.
Time Frame: Baseline up to Day 26
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - 300 mg LY3509754 (Fasted): Participants received a single oral dose of 300 mg LY3509754 under fasting condition.
- Part A - 300 mg LY3509754 (Fed): Participants received a single oral dose of 300 mg LY3509754 under fed condition.
- Part B - Placebo Alone (Day 1): Participants received a single oral dose of placebo on Day 1.
- Part B - Placebo + 200 mg Itraconazole (Day 10): Participants received a single oral dose of placebo and 200 mg itraconazole oral solution on Day 10.
- Part B - 200 mg Itraconazole (Days 4 to 13): Participants received 200 mg itraconazole as an oral solution BID on Day 4 and QD on Days 5 through 13.
- Part B - 10 mg LY3509754 Alone (Day 1): Participants received a single oral dose of 10 mg LY3509754 on Day 1.
- Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10): Participants received a single oral dose of 10 mg LY3509754 and 200 mg itraconazole oral solution on Day 10.
- Part C - 1.2 mg Midazolam (Day -2) [Cohort 2]: Participants received 1.2 mg midazolam as an oral solution on Day -2.
- Part C - Placebo QD (Days 1 to 14) [Cohort 2]: Participants received oral doses of placebo QD for 14 Days upon receiving 1.2 mg midazolam on Day -2.
- Part C - 300 mg LY3509754 QD (Days 1 to 14) [Cohort 2]: Participants received oral doses 300 mg of LY3509754 QD for 14 Days upon receiving 1.2 mg midazolam on Day -2.
- Part C - Placebo QD + 1.2 mg Midazolam (Day 15) [Cohort 2]: Participants received a single oral dose of placebo QD along with 1.2 mg midazolam given as oral solution on Day 15.
- Part C - 300 mg LY3509754 QD + 1.2 mg Midazolam (Day 15) [Cohort 2]: Participants received a single oral dose of 300 mg LY3509754 QD along with 1.2 mg midazolam given as oral solution on Day 15.
Arm/Group | Part A - Placebo (Fasted) | Part A - Placebo (Fed) | Part A - 10 Milligram (mg) LY3509754 (Fasted) | Part A - 30 mg LY3509754 (Fasted) | Part A - 100 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fed) | Part A - 1000 mg LY3509754 (Fasted) | Part A - 2000 mg LY3509754 (Fasted) | Part B - Placebo Alone (Day 1) | Part B - Placebo + 200 mg Itraconazole (Day 10) | Part B - 200 mg Itraconazole (Days 4 to 13) | Part B - 10 mg LY3509754 Alone (Day 1) | Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10) | Part C - Placebo QD [Cohorts 1 and 3] | Part C - 100 mg LY3509754 QD [Cohort 1] | Part C - 1.2 mg Midazolam (Day -2) [Cohort 2] | Part C - Placebo QD (Days 1 to 14) [Cohort 2] | Part C - 300 mg LY3509754 QD (Days 1 to 14) [Cohort 2] | Part C - Placebo QD + 1.2 mg Midazolam (Day 15) [Cohort 2] | Part C - 300 mg LY3509754 QD + 1.2 mg Midazolam (Day 15) [Cohort 2] | Part C - 1000 mg LY3509754 QD [Cohort 3] | Part D (Japanese) - Placebo QD | Part D (Japanese) - 400 mg LY3509754 QD | Part D (Japanese) - 1000 mg LY3509754 QD
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 6 | 9 | 9 | 6 | 6 | 3 | 3 | 11 | 8 | 8 | 4 | 6 | 10 | 2 | 8 | 2 | 8 | 6 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3509754 in Parts A and B
Description: PK: Cmax of LY3509754 in Parts A and B.
Time Frame: Part A: Pre-dose (P), 0.5,1,2,3,4,5,6,8,12,16,24,36,48,72,96 hours (h) post Day 1 dose. Part B: P,0.5,1,2,3,4,6,8,12,16,24,36,48,72,96 h post Day 1 dose; P,0.5,1,2,3,4,6,8,12,16,24,36,48,72,96,120,144,168 h Post Day 10 dose.
Population: All participants who received at least one dose of LY3509754 or itraconazole and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part A - 10 mg LY3509754 (Fasted) | Part A - 30 mg LY3509754 (Fasted) | Part A - 100 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fed) | Part A - 1000 mg LY3509754 (Fasted) | Part A - 2000 mg LY3509754 (Fasted) | Part B - 10 mg LY3509754 Alone (Day 1) | Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10)
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 9 | 6 | 6 | 8 | 8
nanograms per milliliter (ng/mL) | 20.4 (28) | 49.0 (26) | 136 (73) | 384 (62) | 278 (72) | 1390 (55) | 2310 (13) | 15.7 (24) | 43.3 (41)

3. Secondary Outcome: PK: Cmax of LY3509754 in Parts C and D
Description: PK: Cmax of LY3509754 in Parts C and D.
Time Frame: Part C-Cohorts 1 and 3: P,0.5,1,2,3,4,6,8,12,16,24,48,72,96 h Post Day 14 dose. Part C-Cohort 2: P,0.5,1,2,3,4,5,6,8,12,16,24 h Post Day 14 dose. Part D: P,0.5,1,2,3,4,6,8,12,16,24,48,72,96 h Post Day 14 dose.
Population: All participants who received at least one dose of LY3509754 or midazolam and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part C - 300 mg LY3509754 QD (Days 1 to 14) [Cohort 2]: Participants received oral doses of LY3509754 QD for 14 Days upon receiving 1.2 mg midazolam on Day -2.
- Part D(Japanese) - 1000 mg LY3509754 QD: Participants received oral doses of 1000 mg LY3509754 QD for 14 Days.
Arm/Group | Part C - 100 mg LY3509754 QD [Cohort 1] | Part C - 300 mg LY3509754 QD (Days 1 to 14) [Cohort 2] | Part C - 1000 mg LY3509754 QD [Cohort 3] | Part D (Japanese) - 400 mg LY3509754 QD | Part D(Japanese) - 1000 mg LY3509754 QD
Number analyzed (Participants) | 5 | 8 | 6 | 6 | 6
ng/mL | 218 (52) | 458 (50) | 1160 (55) | 805 (30) | 2050 (31)

4. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to 24 Hours Post-dose AUC(0-24) of LY3509754 in Parts A and B
Description: PK: AUC(0-24) of LY3509754 in Parts A and B.
Time Frame: Part A: P, 0.5,1,2,3,4,5,6,8,12,16,24 h post Day 1 dose. Part B: P,0.5,1,2,3,4,6,8,12,16,24 h post Day 1 dose; P,0.5,1,2,3,4,6,8,12,16,24 h Post Day 10 dose.
Population: All participants who received at least one dose of LY3509754 or itraconazole and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram *hour per milliliter (ng*h/mL)
Arm/Group | Part A - 10 mg LY3509754 (Fasted) | Part A - 30 mg LY3509754 (Fasted) | Part A - 100 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fed) | Part A - 1000 mg LY3509754 (Fasted) | Part A - 2000 mg LY3509754 (Fasted) | Part B - 10 mg LY3509754 Alone (Day 1) | Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10)
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 9 | 6 | 6 | 8 | 8
nanogram *hour per milliliter (ng*h/mL) | 153 (20) | 375 (25) | 1340 (60) | 3930 (45) | 2930 (69) | 14900 (42) | 26300 (29) | 135 (29) | 596 (33)

5. Secondary Outcome: PK: AUC(0-24) of LY3509754 in Parts C and D
Description: PK: AUC(0-24) of LY3509754 in Parts C and D.
Time Frame: Part C-Cohorts 1 and 3: P,0.5,1,2,3,4,6,8,12,16,24 h Post Day 14 dose. Part C-Cohort 2: P,0.5,1,2,3,4,5,6,8,12,16,24 h Post Day 14 dose. Part D: P,0.5,1,2,3,4,6,8,12,16,24 h Post Day 14 dose.
Population: All participants who received at least one dose of LY3509754 or midazolam and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part C - 100 mg LY3509754 QD [Cohort 1] | Part C - 300 mg LY3509754 QD (Days 1 to 14) [Cohort 2] | Part C - 1000 mg LY3509754 QD [Cohort 3] | Part D (Japanese) - 400 mg LY3509754 QD | Part D (Japanese) - 1000 mg LY3509754 QD
Number analyzed (Participants) | 5 | 8 | 6 | 6 | 6
ng*h/mL | 2170 (41) | 4050 (38) | 12200 (42) | 7560 (30) | 18000 (22)

ADVERSE EVENTS:
Time Frame: Baseline to Up To Day 26
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Part C - 300 mg LY3509754 QD (Days 1 to 14) [Cohort 2]: Participants received oral doses of 300 mg LY3509754 QD for 14 Days upon receiving 1.2 mg midazolam on Day -2.
- Part D (Japanese) - Placebo QD: Participants received oral doses of placebo QD for 15 Days.
- Part D (Japanese) - 400 mg LY3509754 QD: Participants received oral doses of 400 mg LY3509754 QD for 15 Days.
- Part D (Japanese) - 1000 mg LY3509754 QD: Participants received oral doses of 1000 mg LY3509754 QD for 15 Days.
Arm/Group | Part A - Placebo (Fasted) | Part A - Placebo (Fed) | Part A - 10 Milligram (mg) LY3509754 (Fasted) | Part A - 30 mg LY3509754 (Fasted) | Part A - 100 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fasted) | Part A - 300 mg LY3509754 (Fed) | Part A - 1000 mg LY3509754 (Fasted) | Part A - 2000 mg LY3509754 (Fasted) | Part B - Placebo Alone (Day 1) | Part B - Placebo + 200 mg Itraconazole (Day 10) | Part B - 200 mg Itraconazole (Days 4 to 13) | Part B - 10 mg LY3509754 Alone (Day 1) | Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10) | Part C - Placebo QD [Cohorts 1 and 3] | Part C - 100 mg LY3509754 QD [Cohort 1] | Part C - 1.2 mg Midazolam (Day -2) [Cohort 2] | Part C - Placebo QD (Days 1 to 14) [Cohort 2] | Part C - 300 mg LY3509754 QD (Days 1 to 14) [Cohort 2] | Part C - Placebo QD + 1.2 mg Midazolam (Day 15) [Cohort 2] | Part C - 300 mg LY3509754 QD + 1.2 mg Midazolam (Day 15) [Cohort 2] | Part C - 1000 mg LY3509754 QD [Cohort 3] | Part D (Japanese) - Placebo QD | Part D (Japanese) - 400 mg LY3509754 QD | Part D (Japanese) - 1000 mg LY3509754 QD
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/6 | 0/6 | 0/3 | 0/3 | 0/11 | 0/8 | 0/8 | 0/4 | 0/6 | 0/10 | 0/2 | 0/8 | 0/2 | 0/8 | 0/6 | 0/4 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/2 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/6 | 0/6 | 0/3 | 0/3 | 0/11 | 0/8 | 0/8 | 0/4 | 0/6 | 0/10 | 0/2 | 0/8 | 0/2 | 0/8 | 0/6 | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 1/2 | 0/6 | 1/6 | 0/6 | 0/9 | 2/9 | 0/6 | 0/6 | 0/3 | 0/3 | 4/11 | 0/8 | 1/8 | 1/4 | 2/6 | 1/10 | 0/2 | 2/8 | 1/2 | 0/8 | 2/6 | 2/4 | 4/6 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A - Placebo (Fasted) (N=10) | Part A - Placebo (Fed) (N=2) | Part A - 10 Milligram (mg) LY3509754 (Fasted) (N=6) | Part A - 30 mg LY3509754 (Fasted) (N=6) | Part A - 100 mg LY3509754 (Fasted) (N=6) | Part A - 300 mg LY3509754 (Fasted) (N=9) | Part A - 300 mg LY3509754 (Fed) (N=9) | Part A - 1000 mg LY3509754 (Fasted) (N=6) | Part A - 2000 mg LY3509754 (Fasted) (N=6) | Part B - Placebo Alone (Day 1) (N=3) | Part B - Placebo + 200 mg Itraconazole (Day 10) (N=3) | Part B - 200 mg Itraconazole (Days 4 to 13) (N=11) | Part B - 10 mg LY3509754 Alone (Day 1) (N=8) | Part B - 10 mg LY3509754 + 200 mg Itraconazole (Day 10) (N=8) | Part C - Placebo QD [Cohorts 1 and 3] (N=4) | Part C - 100 mg LY3509754 QD [Cohort 1] (N=6) | Part C - 1.2 mg Midazolam (Day -2) [Cohort 2] (N=10) | Part C - Placebo QD (Days 1 to 14) [Cohort 2] (N=2) | Part C - 300 mg LY3509754 QD (Days 1 to 14) [Cohort 2] (N=8) | Part C - Placebo QD + 1.2 mg Midazolam (Day 15) [Cohort 2] (N=2) | Part C - 300 mg LY3509754 QD + 1.2 mg Midazolam (Day 15) [Cohort 2] (N=8) | Part C - 1000 mg LY3509754 QD [Cohort 3] (N=6) | Part D (Japanese) - Placebo QD (N=4) | Part D (Japanese) - 400 mg LY3509754 QD (N=6) | Part D (Japanese) - 1000 mg LY3509754 QD (N=6)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (5) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Saliva altered (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza b virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/3 (0) | 0/0 (0) | 0/2 (0) | 0/1 (0) | 0/1 (0) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/2 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/1 (0) | 0/2 (0) | 0/4 (0) | 0/1 (0) | 0/3 (0) | 1/1 (1) | 0/3 (0) | 0/0 (0) | 0/1 (0) | 0/2 (0) | 0/2 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Terminated [Terminated due to safety findings].

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT04586920/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT04586920/SAP_001.pdf